CLINICAL TRIAL: NCT06723392
Title: Asymptomatic Bacteriuria in Pregnancy in Low- and Middle-IncomE Countries: A Randomized Controlled Trial of the Global Network for Women's and Children's Health Research
Brief Title: Asymptomatic Bacteriuria in Pregnancy in Low- and Middle-IncomE Countries
Acronym: ABLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: RTI International (Other); University of Virginia (Other); University of Alabama at Birmingham (Other); Thomas Jefferson University (Other); Columbia University (Other); Boston University (Other); University of Colorado, Denver (Other); University of North Carolina, Chapel Hill (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Kinshasa School of Public Health (Other); Institute of Nutrition of Central America and Panama (Other); Lata Medical Research Foundation, Nagpur (Other); Aga Khan University (Other); University Teaching Hospital, Lusaka, Zambia (Other); KLE Academy of Higher Education and Research (Deemed- to- be-University), Jawaharlal Nehru Medical College (JNMC), Belagavi, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP ABLE
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth; Small for Gestational Age (SGA); Stillbirth; Bacteriuria (Asymptomatic) in Pregnancy
Keywords: asymptomatic bacteriuria; small vulnerable newborn; preterm birth; small for gestational agea; still birth; SVN/SB; oral nitrofurantoin monohydrate/macrocrystals; Global Network; Bangladesh; India; Pakistan; Democratic Republic of Congo; Zambia; Guatemala
MeSH Terms: conditions — Premature Birth; Stillbirth; Bacteriuria | interventions — Nitrofurantoin

STUDY DESIGN:
Intervention Model Description: Parallel-arm, double-blind, placebo-controlled, 2:1 allocation, randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral nitrofurantoin monohydrate/macrocrystals (Experimental): Pregnant individuals with AB randomized to receive a 7-day course of oral NM/M 100 mg twice daily (total of 14 doses)
  Interventions: Drug: Oral nitrofurantoin monohydrate/macrocrystals
- Placebo (Placebo Comparator): Pregnant individuals with AB randomized to a receive a 7-day course of oral placebo 100 mg twice daily (total of 14 doses)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral nitrofurantoin monohydrate/macrocrystals — 7-day course of oral nitrofurantoin monohydrate/macrocrystals 100 mg twice daily (total of 14 doses)
  Arms: Oral nitrofurantoin monohydrate/macrocrystals
Other: Placebo — 7-day course of oral placebo 100 mg twice daily (total of 14 doses)
  Arms: Placebo

SUMMARY:
This study, Asymptomatic Bacteriuria in Pregnancy in Low- and Middle-IncomE Countries (ABLE), is designed as a 2-arm randomized controlled trial (RCT) focused on pregnant individuals and newborn infants. A positive outcome of this study will contribute to global progress toward WHO Sustainable Development Goal Target 3.2 [End preventable deaths of newborns and children under 5 years of age] by examining the potential impact of this practice to reduce the incidence of SVN/SB and the lifelong health consequences associated with SVNs. In addition, the study will further explore the role and potential benefits of antibiotic treatment of AB in the pregnant individual. In total, 1,134 eligible participants, or approximately 162 per research site, will be randomized in the trial by the research teams in each of the seven international sites that, together with their United States of America (US) partners, participate in the Eunice Kennedy Shriver National Institute of Child Health and Human Development's (NICHD's) Global Network for Women's and Children's Health Research (GN).

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet the following criteria are eligible for randomization:

* Enrolled in GN MNHR
* Established pregnancy ≥12 and ≤20 weeks GA by last menstrual period and/or clinical assessment and/or ultrasonography
* Age: 18 years (or lower limit age eligible*) to 49 years

  * Some sites will be able to include individuals giving birth regardless of age if they are considered an adult or an emancipated minor. However, other sites will require individuals to be at least 18 years of age. The investigators will adhere to local regulations.
* Expressed understanding of study procedures and willingness to complete screening, randomization, study drug administration and follow-up
* Able to provide informed consent
* Presence of a single bacterial isolate (>105 colony forming unit (CFU)/mL) in urine at enrollment
* Intent to remain in study area for at least 42 days PP

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible for randomization:

* Gestational age <12 weeks or >20 weeks
* Received treatment with any antibiotic within 14 days before screening visit
* Current symptoms of UTI
* History of allergy to nitrofurantoin
* Pregnancy loss / miscarriage prior to randomization
* Currently taking magnesium-containing antacid
* Any illness / condition (e.g., anemia, diabetes, renal disease, pulmonary disease) requiring immediate medical care per site PI assessment
* Enrollment in another trial that per the study MOP will impact this trial

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1134 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of small vulnerable newborn (SVN) or stillbirth (SB) | From Pregnancy until 42 days postpartum
  SVN/SB, defined by the occurrence of any of the following:
  * PTB, defined by birth <37 completed weeks gestation;
  * SGA, defined by birth weight <10th percentile of weight for gestational age, using INTERGROWTH 21st international, sex-specific birthweight standards; or
  * SB, defined by fetal loss or SB > 22 weeks' gestation.

CONTACTS AND LOCATIONS:
Locations (7):
- Icddr,B, Dhaka, Bangladesh, Bangladesh
- Kinshasa School of Public Health, Kinshasa, DRC, Democratic Republic of the Congo
- Institue for Nutrition of Central America and Panama (INCAP), Guatemala City, Departamento de Guatemala, Guatemala
- India (2):
  - KLE Academy of Higher Education and Research, Belagavi, Karnataka
  - Lata Medical Research Foundation, Nagpur, Maharashtra
- Aga Khan University, Karachi, Pakistan, Pakistan
- University Teaching Hospital, Lusaka, Zambia, Zambia